CLINICAL TRIAL: NCT01444521
Title: Genotype-drive Phase II Study of Novel Irinotecan-Cisplatin Combination as First-line Therapy for Advanced Gastric Cancer
Brief Title: Genotype-drive Study of Irinotecan-Cisplatin Combination for Advanced Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Jing Huang, Principle Investigator, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CH-GI-017
Record Dates: First submitted 2011-09-25; First posted 2011-09-30 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: Gastric Cancer
Keywords: advanced gastric cancer; irinotecan; cisplatin
MeSH Terms: conditions — Stomach Neoplasms | interventions — Irinotecan; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single-arm Irinotecan-Cisplatin (Experimental)
  Interventions: Drug: irinotecan and cisplatin

INTERVENTIONS:
Drug: irinotecan and cisplatin — irinotecan 125 mg/m2 will be administered as an intravenous (IV) infusion over half a hour on Days 1; Cisplatin 60 mg/m2 will be administered as an intravenous (IV) infusion on Days 2, and to take enough hydration in the day and the next day.
  14 days as a cycle, up to 8 cycles.
  Other Names: CAMPT

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of first-line chemotherapy with cisplatin and irinotecan in advanced gastric cancer, and try to find out the optimal dosage of combination chemotherapy.

DETAILED DESCRIPTION:
Open label single arm phase II study of cisplatin and irinotecan in patients with advanced gastric carcinoma not previously treated with palliative chemotherapy. 40 Patients will be enrolled in this local trial. The primary objective of this study is to determine the response rate of the treatment.Schedule for this study is as follows: 8 cycles/14 days of irinotecan 125 mg/m2 on Day 1 and cisplatin 50 mg/m2 on Day2. This study will also include genotype investigations of UGT1A1 and ERCC1 expression in order to assess determinants of efficacy and toxicity of the treatment with cisplatin and irinotecan in the study population.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis of adenocarcinoma of the stomach (including adenocarcinoma of the gastroesophageal junction)
* Stage III or Stage IV disease, according to American Joint Committee on Cancer criteria
* Patients with UGT1A1*28 genotype 6/6 or 6/7
* Performance Status of 0-2 on the Eastern Cooperative Oncology Group (ECOG) performance status Scale
* Previous adjuvant or pre-operative chemotherapy without containing irinotecan or platinum at least 6 months before enrollment
* Adequate organ function including the following:

Bone marrow: absolute neutrophil count (ANC) >or equal to 1.5 * 109/L, platelets >or equal to 100 *109/L, hemoglobin > or equal to 10 g/dL.

Hepatic: bilirubin < or equal to 1.5 x ULN; alkaline phosphatase, aspartate transaminase (AST) and alanine transaminase (ALT) < or equal to 3 x ULN (alkaline phosphatase, AST, ALT minor or equal to 5 x ULN is acceptable if liver has tumor involvement), serum albumin > or equal to3g/dL.

Renal: Calculated creatinine clearance major or equal to 60 ml/min (using the standard Cockcroft-Gault formula).

Exclusion Criteria:

* No Prior palliative chemotherapy for advanced disease
* Previous radiation therapy is allowed but should have been limited and must not have included whole pelvis radiation. Patients must have recovered from the toxic effects of the treatment prior to study enrollment (except for alopecia). Prior radiotherapy must be completed at least 30 days before study enrollment
* Known or suspected brain metastasis
* Second primary malignancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-04; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Overall response rate | 1 year
  The primary objective of this study is to determine the response rate of CPT11 plus cisplatin as first-line therapy in patients with advanced gastric carcinoma.

SECONDARY OUTCOMES:
Time to event efficacy | 1 year
  The secondary objectives of this study are to evaluate:
  The following time to event efficacy measures:
  * Duration of overall response for responding patients
  * Time to documented progressive disease
  * Overall survival
  * The quantitative and qualitative toxicity of irinotecan plus cisplatin.
  * Determinants of efficacy and toxicity of the treatment with irinotecan and cisplatin in the patient population by means of pharmacogenomic investigations: Quantitative analysis of UGT1A1 and ERCC1

CONTACTS AND LOCATIONS:
Overall Officials: Jing Huang, M.D.,Ph.D, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, China

REFERENCES:
- [Result] Koizumi W, Kurihara M, Satoh A, Takiuchi H, Tanabe S, Shimada K, Iwasaki R, Saigenji K. Phase 1/11 study of bi-weekly irinotecan plus cisplatin in the treatment of advanced gastric cancer. Anticancer Res. 2005 Mar-Apr;25(2B):1257-62. PMID 15865075
- [Result] Satoh T, Ura T, Yamada Y, Yamazaki K, Tsujinaka T, Munakata M, Nishina T, Okamura S, Esaki T, Sasaki Y, Koizumi W, Kakeji Y, Ishizuka N, Hyodo I, Sakata Y. Genotype-directed, dose-finding study of irinotecan in cancer patients with UGT1A1*28 and/or UGT1A1*6 polymorphisms. Cancer Sci. 2011 Oct;102(10):1868-73. doi: 10.1111/j.1349-7006.2011.02030.x. Epub 2011 Aug 12. PMID 21740478